CLINICAL TRIAL: NCT00166348
Title: Efficacy of Group Based Cognitive Rehabilitation Following Acquired Brain Injury
Brief Title: Does Cognitive Rehabilitation Demonstrate Benefits in the Group Setting With People Whom Have Experienced Brain Injury?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Nicloe Holzworth, OTR/L (Unknown); Bergequist, Thomas, Ph.D. (Individual); Brown, Allen, M.D. (Individual); Sue Lepore, OTR/L (Unknown); Walter Stobaugh. LICSW (Unknown)
Responsible Party: Merri L Vitse, AS, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1069-03
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Brain Injuries
Keywords: Cognitive Rehabilitation
MeSH Terms: conditions — Brain Injuries

INTERVENTIONS:
Behavioral: Cognitive Group Therapy

SUMMARY:
The purpose of this study is to determine whether there is benefit from providing cognitive rehabilitation in the group setting. Several standardized tools will be used to measure progress when a participant enters the group, leaves the group and at a one year follow-up.

DETAILED DESCRIPTION:
This research study will look at the outcome benefits of providing cognitive rehabilitation, utilizing the group process. Criteria for selecting the appropriate participants, group format and structure, as well as use of standardized assessments. The assessments used: Three Step Calendar Approach, (Sohlberg and Mateer) Satisfaction With Life scale (SWLS), Community Integration Questionnaire (CIQ), Independent Living Scale, and the Vocational Independence Scale. The group setting provides an atmosphere to work on building communication skills through peer feedback and to develop psychological coping strategies. Techniques such as the problem solving format and a calendar system. Analysis and outcomes of 17 past group participants were analyzed supporting cognitive rehabilitation in the group setting.

Of the 20 participants, 3 chose not to be included.

ELIGIBILITY:
Inclusion Criteria:

* All participants involved in the Cognitive Rehabilitation Outpatient Group within the study time frame are eligible to be in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-03; Primary Completion 2007-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
provide evidence which supports cognitive therapy in a group setting
less labor intensive
cost effectiveness
peer feedback is effective

CONTACTS AND LOCATIONS:
Overall Officials: Merri L Vitse, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States